CLINICAL TRIAL: NCT04565158
Title: Assessment of Sleep Disruption in Women With Bilateral Salpingo-Oophorectomy - A SCORE Ancillary Study
Brief Title: Sleep in Women With Bilateral Salpingo-Oophorectomy
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Naima Covassin, Principal Investigator, Mayo Clinic
Other Study IDs: 20-005982
Record Dates: First submitted 2020-08-31; First posted 2020-09-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Bilateral Salpingo-oophorectomy
Keywords: salpingo-oophorectomy; sleep; cognitive decline
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with bilateral salpingo-oophorectomy (BSO)
- Women without bilateral salpingo-oophorectomy (BSO)

SUMMARY:
The purpose of this research study is the compare objective and subjective sleep characteristics in women who have undergone removal of both ovaries (bilateral salpingo-oophorectomy) before natural menopause compared to women who did not undergo this procedure.

ELIGIBILITY:
Inclusion Criteria:

* Women who participate in the parent SCORE studies (NCT03821857)

Exclusion Criteria:

* Night shift workers will be excluded

Min Age: 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cases: Women who underwent bilateral salpingo-oophorectomy prior to natural menopause Controls: Women who did not undergo bilateral salpingo-oophorectomy prior to natural menopause
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-11-06 (Actual)

PRIMARY OUTCOMES:
prevalence of sleep disorders | 2 years
  prevalence of sleep disordered breathing, insomnia, and restless legs syndrome
prevalence of short sleep duration | 2 years
  objective sleep duration from actigraphy/polysomnography and subjective sleep duration from self-report
prevalence of poor sleep quality | 2 years
  objective sleep quality from actigraphy/polysomnography and subjective sleep quality from self-report

OTHER OUTCOMES:
exploratory correlation between sleep measures and cognitive function | 2 years
  correlation between objective and subjective sleep measures (sleep duration, sleep quality and sleep disorders) and tests of cognitive function (attention, memory, language, and global cognitive function)
exploratory correlation between sleep measures and neuroimaging | 2 years
  correlation between objective and subjective sleep measures (sleep duration, sleep quality and sleep disorders) and tests of cognitive function (attention, memory, language, and global cognitive function)

CONTACTS AND LOCATIONS:
Overall Officials: Naima Covassin, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials